CLINICAL TRIAL: NCT02495922
Title: A Randomized Phase III Trial on the Effect of Elotuzumab in VRD Induction /Consolidation and Lenalidomide Maintenance in Patients With Newly Diagnosed Myeloma
Brief Title: A Phase III Trial on the Effect of Elotuzumab in VRD Induction /Consolidation and Lenalidomide Maintenance in Patients With Newly Diagnosed Myeloma
Acronym: GMMG-HD6
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Heidelberg Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Goldschmidt, Prof. Dr., University of Heidelberg Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMMG HD6
Record Dates: First submitted 2015-06-24; First posted 2015-07-13 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1 (Active Comparator): Induction therapy with 4 cycles VRD (Velcade, Revlimid, Dexamethasone), 21 days per cycle, intensification (mobilization and autologous stem cell transplantation), consolidation therapy with 2 cycles VRD (Velcade, Revlimid, Dexamethasone), 21 days per cycle. Maintenance therapy: 26 cycles (28 days) with lenalidomide (Dexamethasone on day 1 and 15 in cycles 1-6 and on day 1 in cycles 7 to 26).
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone
- A2 (Experimental): Induction therapy with 4 cycles VRD (Velcade, Revlimid, Dexamethasone) 21 days per cycle, intensification (mobilization and autologous stem cell transplantation), consolidation therapy with 2 cycles VRD (Velcade, Revlimid, Dexamethasone) + elotuzumab, 21 days per cycle. Maintenance therapy: 26 cycles (28 days) with lenalidomide + elotuzumab (Dexamethasone on day 1 and 15 in cycles 1-6 and on day 1 in cycles 7 to 26).
  Interventions: Drug: elotuzumab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone
- B1 (Experimental): Induction therapy with 4 cycles VRD (Velcade, Revlimid, Dexamethasone) + elotuzumab , 21 days per cycle, intensification (mobilization and autologous stem cell transplantation), consolidation therapy with 2 cycles VRD (Velcade, Revlimid, Dexamethasone) 21 days per cycle. Maintenance therapy: 26 cycles (28 days) with lenalidomide (Dexamethasone on day 1 and 15 in cycles 1-6 and on day 1 in cycles 7 to 26).
  Interventions: Drug: elotuzumab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone
- B2 (Experimental): Induction therapy with 4 cycles VRD (Velcade, Revlimid, Dexamethasone) + elotuzumab, 21 days per cycle, intensification (mobilization and autologous stem cell transplantation), consolidation therapy with 2 cycles VRD (Velcade, Revlimid, Dexamethasone) + elotuzumab, 21 days per cycle. Maintenance therapy: 26 cycles (28 days) with lenalidomide + elotuzumab (Dexamethasone on day 1 and 15 in cycles 1-6 and on day 1 in cycles 7 to 26).
  Interventions: Drug: elotuzumab; Drug: Lenalidomide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: elotuzumab — 10 mg/kg in the vein( i.v) on day 1,8 and 15 in induction cycle 1 and 2, on day 1 and 11 in induction cycle 3 and 4 (Arm B1 and B2). 10 mg/kg i.v. on day 1,8 and 15 in consolidation cycle 1 and 2 (Arm A2 and B2), 10 mg/kg i.v. on day 1 and15 in maintenance cycle 1-6, 10 mg/kg i.v. on day 1 in maintenance cycle 7-26 (Arm A2 and B2)
  Arms: A2; B1; B2
Drug: Lenalidomide — 25 mg per os on day 1-14 in induction cycle 1-4, 25 mg p.o. on day 1-14 in consolidation cycle 1 and 2, 10 mg p.o. on day 1-28 in maintenance cycle 1-3, 15 mg p.o. on day 1-28 in maintenance cycle 4-26 (all arms)
  Other Names: Revlimid
Drug: Bortezomib — all arms: 1,3 mg/m^2 subcutaneous on day 1, 4, 8 and 11 in 4 induction cycles, 1,3 mg/m^2 subcutaneous on day 1, 8 and 15 in 2 cycles of consolidation
  Other Names: Velcade
Drug: Dexamethasone — 20 mg per os on day 1,2 and 4,5 and 8,9 and 11,12 and 15 in induction cycles 1 and 2. 20 mg per os on day 1,2 and 4,5 and 8,9 and 11,12 in induction cycles 3 and 4 (Arms A1 and A2).
  8 mg per os and 12 mg i.v. on day 1, 8 and 15 and 20 mg per os on days 2,4,5, 9, 11 and 12 in induction cycles 1 and 2. 8 mg per os and 12 mg i.v. on day 1, and 11, 20 mg per os on days 2,4,5,8, 9, and 12 in induction cycles 3 and 4 (Arms B1 and B2).
  20 mg per os on days 1,2, 8,9, 15 and 16 in both cycles of consolidation (Arms A1 and B1). 8 mg per os and 12 mg i.v. on days 1, 8 and 15 and 20 mg per os on days 2, 9 and 16 in both consolidation cycles (Arms A2 and B2).
  12 mg per os on day 1 and 15 in maintenance cycles 1-6, 12 mg per os on day 1 of maintenance cycles 7 and following (Arms A1 and B1). 4 mg per os and 8 mg i.v. on day 1 and 15 in maintenance cycles 1-6, 4 mg per os and 8 mg i.v. on day 1 of maintenance cycles 7 and following (Arms A2 and B2).

SUMMARY:
Trial in patients with newly diagnosed myeloma to evaluate the effect of elotuzumab in induction and consolidation therapy with bortezomib/lenalidomide/dexamethasone and in lenalidomide maintenance treatment

DETAILED DESCRIPTION:
Prospective, multicentre, randomised, parallel group, open, phase III clinical trial, for patients with confirmed diagnosis of untreated multiple myeloma requiring systemic therapy .

Investigational Medicinal Products:Elotuzumab, lenalidomide

Patients are randomized in one of 4 study arms (A1, A2, B1, B2). Patients randomized in arm A1 or A2 will receive 4 cycles VRD (Bortezomib (Velcade®), Lenalidomide (Revlimid®), Dexamethasone). Patients in arm B1 or B2 will additionally receive the monoclonal antibody Elotuzumab in the 4 cycles VRD. After induction therapy patients undergo intensifying therapy according to GMMG standard (usually mobilization therapy followed by stem cell collection and autologous stem cell transplantation). After intensification a consolidation therapy will be performed with two cycles VRD (A1 und B1) or VRD+ Elotuzumab (A2 und B2), followed by Lenalidomide maintenance therapy with (arm A2 and B2) or without (arm A1 and B1) additional Elotuzumab. Maintenance therapy will be performed for 2 years.

Primary objective is the determination of the best of four treatment strategies regarding progression-free survival (PFS), defined as time from randomisation to progression or death from any cause whichever occurs first.

The duration of the trial for each patients is expected to be 36-39 months (induction and intensification treatment: 7-10 months, 3 months rest between intensification and start of consolidation, consolidation 2 months, maintenance phase 24 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting all of the following criteria will be considered for admission to the trial:
* Confirmed diagnosis of untreated multiple myeloma requiring systemic therapy (diagnostic criteria (IMWG updated criteria (2014) )
* Measurable disease, defined as any quantifiable monoclonal protein value, defined by at least one of the following three measurements:

  * Serum M-protein ≥ 10g/l (for IgA ≥ 5g/l)
  * Urine light-chain (M-protein) of ≥ 200 mg/24 hours
  * Serum FLC assay: involved FLC level ≥ 10 mg/dl provided sFLC ratio is abnormal
* Age 18 - 70 years inclusive
* WHO performance status 0-3 (WHO=3 is allowed only if caused by MM and not by co-morbid conditions)
* Negative pregnancy test at inclusion (women of childbearing potential)
* For all men and women of childbearing potential: patients must be willing and capable to use adequate contraception during the complete therapy. Patients must agree on the requirements regarding the lenalidomide pregnancy prevention programme described in chapter 6.
* All patients must

  * agree to abstain from donating blood while taking lenalidomide and for 28 days following discontinuation of lenalidomide therapy
  * agree not to share study drug lenalidomide with another person and to return all unused study drug to the investigator or pharmacist
* Ability of patient to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrollment in the trial)

Exclusion Criteria:

* Patients presenting with any of the following criteria will not be included in the trial:
* Patient has known hypersensitivity to any drugs given in the protocol, notably bortezomib, lenalidomide, dexamethasone and elotuzumab or to any of the constituent compounds (incl. boron and mannitol).
* Systemic AL amyloidosis (except for AL amyloidosis of the skin or the bone marrow)
* Previous chemotherapy or radiotherapy during the past 5 years except local radiotherapy in case of local myeloma progression.
* Severe cardiac dysfunction (NYHA classification III-IV)
* Significant hepatic dysfunction (serum bilirubin ≥ 1,8mg/dl and/or ASAT and/or ALAT ≥ 2.5 times normal level), unless related to myeloma.
* Patients with renal insufficiency requiring hemodialysis
* HIV positivity
* Patients with active or history of hepatitis B or C
* Patients with active, uncontrolled infections
* Patients with peripheral neuropathy or neuropathic pain, CTC grade 2 or higher (as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0)
* Patients with a history of active malignancy during the past 5 years with the exception of basal cell carcinoma of the skin or stage 0 cervical carcinoma treated with curative intent
* Patients with acute diffuse infiltrative pulmonary and/or pericardial disease
* Autoimmune hemolytic anemia with positive Coombs test or immune thrombocytopenia
* Platelet count < 75 x 109/l, or, dependent on bone marrow infiltration by plasma cells, platelet count < 30 x 109/l (patients with platelet count < 75 x 109/l, but > 30 x 109/l may be eligible if percentage of plasma cells in bone marrow is ≥ 50%), (transfusion support within 14 days before the test is not allowed)
* Haemoglobin ≤ 8.0 g/dl, unless related to myeloma
* Absolute neutrophil count (ANC) < 1.0 x 10^9/l (the use of colony stimulating factors within 14 days before the test is not allowed), unless related to myeloma
* Pregnancy and lactation
* Participation in other clinical trials. This does not include long-term follow-up periods without active drug treatment of previous studies during the last 6 months.

No patients will be allowed to enrol in this trial more than once.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2015-06; Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
the best of four treatment strategies regarding Progression Free Survival (PFS) | time from randomization to progression or death from any cause whichever comes first, censored after two years of maintenance therapy (i.e. approx. after 36 months after randomisation)
  response evaluation

SECONDARY OUTCOMES:
overall survival | time from randomisation to time of death from any cause. Patients still being alive at the time of the analysis will be censored at the date last known to be alive. (assessed up to 80 months)
  survival status
complete response rates after induction | approx. after 3 months (after induction therapy)
  response evaluation
complete response rates after consolidation | approx. after 9 months (after consolidation therapy)
  response evaluation
Progression Free Survival after end of trial | time from randomisation to progression or death from any cause whichever comes first, censored at the end date of the trial (i.e. assessed up to 80 months)
  response evaluation
best response to treatment during the study | response assessment after ca. 3 months, 4 months, 7 months, 9 months,11 months, 14 months, and subsequently every 3 months during maintenance treatment, up to 35 months after start of study treatment.
  response evaluation
time to progression, censored at end of the trial | From date of randomization until the date of first documented progression, assessed up to 80 months
  Response evaluation
duration of response, censored at end of the trial | assessed up to 80 months
  response evaluation
toxicity during induction treatment, consolidation and maintenance treatment with respect to adverse Events of CTCAE grade 3 or higher | from first administration of study drug until 40 days after last administration of study drug or any drug of the study treatment or upon start of a new subsequent chemotherapy, whichever occurs first
  toxicity according CTCAE Version 4.0
Quality of Life assessment | assessed at baseline, after ca. 3 months, 7 months, 9 months, subsequently every 6 months, up to 36 months
  Questionnaires EORTC-QLQC30 and EORTC-QLQMY20

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Goldschmidt, Prof. Dr., Principal Investigator — Med. Klinik V, University Hospital Heidelberg
Locations (68):
- Germany (68):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - MVZ Onkologie gGmbH der Klinikum Mittelbaden gGmbH, Baden-Baden
  - HELIOS Klinikum, Klinik für Hämatologie, Onkologie und Immunologie, Berlin
  - Onkologisches MVZ Berlin Tegel, Berlin
  - Charité Campus Benjamin Franklin, III. Med. Abt. (Hämatologie/Onkologie), Berlin
  - Klinikum Bielefeld, Klinik für Hämatologie, Onkologie und Palliativmedizin, Bielefeld
  - Studiengesellschaft Onkologie Bielefeld GbR, Bielefeld
  - Hämatologisch-onkologische Schwerpunktpraxis, Bochum
  - Medizinische Universitätsklinik, Knappschaftskrankenhaus, Bochum
  - Universitätsklinikum Bonn, Medizinische Klinik und Poliklinik III, Schwerpunkt Onkologie, Hämatologie und Rheumatologie, Bonn
  - ZAHO, Zentrum für ambulante Hämatologie und Onkologie, Bonn
  - Schwerpunktpraxis für Onkologie/Hämatologie, Bottrop
  - Klinikum Chemnitz GmbH, Innere Medizin III, Chemnitz
  - Universitätsklinikum Köln, Klinik I - Innere Medizin, Cologne
  - Onkologisches Studienzentrum Darmstadt, Darmstadt
  - Klinikum Darmstadt, Med. Klinik V, Hämatologie/Onkologie, Darmstadt
  - HELIOS St. Johannes Klinik, Akademisches Krankenhaus der Heinrich-Heine-Universität Düsseldorf, Duisburg
  - MVZ Düsseldorf GmbH, Düsseldorf
  - Sana Kliniken Düsseldorf GmbH, Düsseldorf
  - Universitätsklinikum Düsseldorf, Klinik für Hämatologie,Onkologie und Klin. Immunologie, Düsseldorf
  - Universitätsklinik Erlangen, Erlangen
  - St.-Antonius-Hospital Klinik f. Hämatologie und Onkologie, Eschweiler
  - Universitätsklinikum Essen, Klinik für Hämatologie, Essen
  - Ev. Krankenhaus Essen-Werden gGmbH, Zentrum für Innere Medizin, Klinik für Hämatologie, Onkologie und Stammzelltransplantation, Essen
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Universitätsklinikum Frankfurt, Goethe-Universität Medizinische Klinik II, Frankfurt am Main
  - Praxis und Tagesklinik Friedrichshafen, Friedrichshafen
  - Gemeinschaftspraxis Schmitt/Eulenbuch, Gerlingen
  - Justus-Liebig-Universität, Medizinische Klinik IV, Giessen
  - Kath. Krankenhaus Hagen gGmbH, Abt. Hämatologie/Onkologie, Hagen
  - Universitätsklinikum Hamburg-Eppendorf, II - Med. Klinik und Poliklinik, Hamburg
  - Asklepios Klinik Hamburg Altona, II. Med. Klinik, Hamburg
  - Evangelisches Krankhaus Hamm gGmbH, Hamm
  - Onkologische Schwerpunktpraxis, Heidelberg
  - University Hospital Heidelberg, Med. Klinik V, Heidelberg
  - Onkologische Schwerpunktpraxis, Heilbronn
  - SLK Kliniken Heilbronn, Med. Klinik III, Heilbronn
  - Universitätsklinikum des Saarlandes, Innere Medizin I, Homburg
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Onkologische Schwerpunktpraxis Karlsruhe, Karlsruhe
  - Onkologische Gemeinschaftspraxis Kassel, Kassel
  - Praxisklinik für Hämatologie und Onkologie, Koblenz
  - Onkologisches Zentrum, Gemeinschaftspraxis f. Hämatologie u. Onkologie im Caritas KH, Lebach
  - Klinikum Lippe GmbH, Hämatologie-Onkologie, Lemgo
  - Schwerpunktpraxis für Hämatologie und Onkologie, Ludwigsburg
  - Med. Klinik A, Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen am Rhein
  - Internistische Schwerpunktpraxis für Hämatologie und Onkologie, Mainz
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, III. Med. Klinik, Mainz
  - III. Medizinische Klinik Hämatologie und Internistische Onkologie, Mannheim
  - Mannheimer Onkologie Praxis, Mannheim
  - Philipps-Universität Marburg, Hämatologie/Onkologie/Immunologie, Marburg
  - Mühlenkreiskliniken (AöR) Johannes Wesling Klinikum Minden, Hämatologie/Onkologie, Hämostaseologie und Palliativmedizin, Minden
  - Krankenhaus Maria Hilf GmbH, Franziskuskrankenhaus, Med. Klinik I, Mönchengladbach
  - Praxis für Hämatologie und internistische Onkologie, Oberhausen
  - Internistisch, Onkologische Gemeinschaftspraxis Dres. Balló, Offenbach
  - Onkologische Praxis Oldenburg, Oldenburg
  - Krankenhaus Barmherzige Brüder, Klinik für Onkologie und Hämatologie, Regensburg
  - Klinikum am Steinenberg, Ermstalklinik, Medizinische Klinik I, Reutlingen
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Innere Medizin III, Schwäbisch Hall
  - ZAHO-Zentrum für ambulante Hämatologie und Onkologie, Standort Siegburg, Siegburg
  - Diakonie Klinikum Jung-Stilling-Krankenhaus, Medizinische Klinik, Siegen
  - Onkologische Schwerpunktpraxis für Onkologie und Gastroenterologie, Singen
  - Onkologische Schwerpunktpraxis Speyer, Speyer
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - University Hospital Tübingen, Med. Klinik und Poliklinik, Abt. II, Tübingen
  - Schwarzwald-Baar Klinikum, Klinik für Innere Medizin II, Villingen-Schwenningen
  - Rems-Murr-Klinikum gGmbH Winnenden, Winnenden

REFERENCES:
- [Derived] Mai EK, Goldschmid H, Miah K, Bertsch U, Besemer B, Hanel M, Krzykalla J, Fenk R, Schlenzka J, Munder M, Durig J, Blau IW, Huhn S, Hose D, Jauch A, Kunz C, Mann C, Weinhold N, Scheid C, Schroers R, von Metzler I, Schieferdecker A, Thomalla J, Reimer P, Mahlberg R, Graeven U, Kremers S, Martens UM, Kunz C, Hensel M, Benner A, Seidel-Glatzer A, Weisel KC, Raab MS, Salwender HJ; German-speaking Myeloma Multicenter Group (GMMG) HD6 investigators. Elotuzumab, lenalidomide, bortezomib, dexamethasone, and autologous haematopoietic stem-cell transplantation for newly diagnosed multiple myeloma (GMMG-HD6): results from a randomised, phase 3 trial. Lancet Haematol. 2024 Feb;11(2):e101-e113. doi: 10.1016/S2352-3026(23)00366-6. PMID 38302221
- [Derived] Maura F, Rajanna AR, Ziccheddu B, Poos AM, Derkach A, Maclachlan K, Durante M, Diamond B, Papadimitriou M, Davies F, Boyle EM, Walker B, Hultcrantz M, Silva A, Hampton O, Teer JK, Siegel EM, Bolli N, Jackson GH, Kaiser M, Pawlyn C, Cook G, Kazandjian D, Stein C, Chesi M, Bergsagel L, Mai EK, Goldschmidt H, Weisel KC, Fenk R, Raab MS, Van Rhee F, Usmani S, Shain KH, Weinhold N, Morgan G, Landgren O. Genomic Classification and Individualized Prognosis in Multiple Myeloma. J Clin Oncol. 2024 Apr 10;42(11):1229-1240. doi: 10.1200/JCO.23.01277. Epub 2024 Jan 9. PMID 38194610
- [Derived] Kauer J, Freundt EP, Schmitt A, Weinhold N, Mai EK, Muller-Tidow C, Goldschmidt H, Raab MS, Kriegsmann K, Sauer S. Stem cell collection after lenalidomide, bortezomib and dexamethasone plus elotuzumab or isatuximab in newly diagnosed multiple myeloma patients: a single centre experience from the GMMG-HD6 and -HD7 trials. BMC Cancer. 2023 Nov 21;23(1):1132. doi: 10.1186/s12885-023-11507-9. PMID 37990162
- [Derived] Salwender H, Bertsch U, Weisel K, Duerig J, Kunz C, Benner A, Blau IW, Raab MS, Hillengass J, Hose D, Huhn S, Hundemer M, Andrulis M, Jauch A, Seidel-Glaetzer A, Lindemann HW, Hensel M, Fronhoffs S, Martens U, Hansen T, Wattad M, Graeven U, Munder M, Fenk R, Haenel M, Scheid C, Goldschmidt H. Rationale and design of the German-speaking myeloma multicenter group (GMMG) trial HD6: a randomized phase III trial on the effect of elotuzumab in VRD induction/consolidation and lenalidomide maintenance in patients with newly diagnosed myeloma. BMC Cancer. 2019 May 28;19(1):504. doi: 10.1186/s12885-019-5600-x. PMID 31138244